CLINICAL TRIAL: NCT03051997
Title: Behavioral Incentives to Increase Caregiver Engagement in Juvenile Drug Courts
Brief Title: Increasing Caregiver Engagement in Juvenile Drug Courts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Wayne State University (Other); Alliant International University (Other); Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MD011322 (NIH); R01MD011322 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver Contingency Management + Usual Drug Court Treatment (Experimental): This group will receive a caregiver contingency management intervention plus the standard outpatient substance abuse treatment services provided at JDC.
  Interventions: Behavioral: Caregiver Contingency Management + Usual Drug Court Treatment
- Usual Drug Court Treatment (Active Comparator): This group will receive the standard outpatient substance abuse treatment services provided at JDC.
  Interventions: Behavioral: Usual Drug Court Treatment

INTERVENTIONS:
Behavioral: Caregiver Contingency Management + Usual Drug Court Treatment — In addition to receiving JDC treatment as usual described below, caregiver participants will receive prize draws for engaging in activities consistent with their adolescents' successful completion of the JDC program during the time the youth is actively involved in JDC and substance abuse treatment. Specific activities that may be reinforced include: attendance at drug court hearings; accompanying the youth to probation meetings; participating in home visits; attendance at the youth's drug treatment sessions; attendance at mental health provider meetings; attending groups for parents of youth with substance abuse issues; and completing other verifiable treatment-related activities. All activities will meet the goals of (directly or indirectly) enhancing caregiver participation in the JDC and/or treatment process. Caregivers will receive escalating chances for tangible reinforcers each week for completing up to 3 of the activities agreed upon by the caregiver and the therapist.
  Arms: Caregiver Contingency Management + Usual Drug Court Treatment
Behavioral: Usual Drug Court Treatment — Standard outpatient substance abuse treatment services that a young person would receive while participating in JDC.
  Arms: Usual Drug Court Treatment

SUMMARY:
The purpose of this study is to test a prize-based contingency management intervention for increasing caregiver engagement in juvenile drug court and adolescent drug treatment, and for achieving the ultimate outcomes of reduced substance use and delinquent behavior among drug court-involved youth.

DETAILED DESCRIPTION:
Juvenile offenders with substance abuse problems represent a large and underserved population that is at high risk of deleterious outcomes and long-term costs for themselves, their families, communities, and society. Moreover, a high percentage of substance abusing adolescents continue to abuse substances and engage in criminal activity into adulthood. Although one juvenile justice intervention, Juvenile Drug Court (JDC), has emerged as a promising model for reducing drug use and delinquency among youth, its effectiveness is variable. Drug court outcomes may be compromised by the lack of caregiver engagement in JDC processes and adolescent drug treatment. Incorporating easily implemented evidence-based incentive programs in JDCs might improve their effectiveness in reducing youth drug use and re-offending. An extensive body of research supports the critical role that families play in the etiology, maintenance, and treatment of adolescent substance abuse. Although family-based interventions for adolescent substance abuse have been shown to be superior to other treatment modalities, parents must attend treatment and participate in meaningful ways for these superior outcomes to be realized. This randomized clinical trial will examine the efficacy of a prize-based contingency management intervention for increasing caregiver engagement (attendance and participation) in JDC and adolescent drug treatment. This caregiver contingency management intervention (CCM) will be compared with drug court treatment as usual (TAU). Increased caregiver participation is predicted to improve adolescent outcomes (decreased drug use and delinquent behavior). One hundred and eighty youth enrolled in JDC will be randomly assigned along with a parent/caregiver to TAU or CCM. Analyses will examine measures of caregiver engagement in JDC as well as youth substance use (urine drug screens) and delinquent activity. Results from this study will demonstrate the effectiveness of CCM procedures for increasing caregiver attendance and participation in JDC and adolescent drug treatment above and beyond drug court and usual care. If effective, the CCM approach may ultimately be used to enhance JDC outcomes, thereby reducing substance use and recidivism in juvenile offenders served by this promising juvenile justice intervention.

ELIGIBILITY:
Inclusion Criteria for youth:

* Involved in juvenile drug court
* Aged 13-17 years
* Youth is willing to participate
* At least one caregiver is willing to participate in the youth's treatment
* Fluent in English or Spanish

Exclusion Criteria for youth:

* Diagnosed with intellectual disability or autism spectrum disorder

Inclusion Criteria for caregivers:

* Caregiver of youth involved in juvenile drug court
* Caregiver is willing to participate
* Fluent in English or Spanish

Exclusion Criteria for caregivers:

* Diagnosed with intellectual disability or autism spectrum disorder

Inclusion Criteria for therapists:

* Providing substance abuse treatment to a youth in juvenile drug court

Exclusion Criteria for therapists:

* None

Inclusion Criteria for Juvenile Drug Court Personnel:

* Personnel working in juvenile drug court

Exclusion Criteria for Juvenile Drug Court Personnel:

* None

Ages: 13 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe Cunningham, Ph.D., Principal Investigator — Medical University of South Carolina; David Ledgerwood, Ph.D., Principal Investigator — Wayne State University; Stacy Ryan, Ph.D., Study Director — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Montgomer County Juvenile Court, 380 West Second Street, Dayton, Ohio
  - Nueces County Juvenile Court/Juvenile Treatment Court, Corpus Christi, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledgerwood DM, Cunningham PB. Juvenile Drug Treatment Court. Pediatr Clin North Am. 2019 Dec;66(6):1193-1202. doi: 10.1016/j.pcl.2019.08.011. PMID 31679607

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled adolescent-caregiver dyads. The reported enrollment (n=53) reflects dyads. Outcome and adverse event data were collected only for adolescents unless otherwise noted. Counts represent dyads. Individual counts for adolescents and caregivers were not separately tracked for milestones.
Period: Overall Study
Arm/Group | Caregiver Contingency Management + Usual Drug Court Treatment | Usual Drug Court Treatment
Started | 32 | 21
Completed | 32 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Measures were only collected for adolescents participants. They were not collected for Caregivers
Groups:
- Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents): This group will receive a caregiver contingency management intervention plus the standard outpatient substance abuse treatment services provided at JDC.
  Baseline Measures is for the adolescent participants
- Usual Drug Court Treatment (Adolescents): This group will receive the standard outpatient substance abuse treatment services provided at JDC.
  Baseline Measures is for the adolescent participants
- Total: Total of all reporting groups
Arm/Group | Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents) | Usual Drug Court Treatment (Adolescents) | Total
Number analyzed (Participants) | 32 | 21 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.46 (1.40) | 15.46 (1.40) | 15.46 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 14
  Male | 21 | 18 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 5 | 16
  White | 17 | 10 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 32 | 21 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Urine Drug Screens at 5 Months Post-baseline
Description: This measure reflects the number of positive urine drug screens for THC, amphetamines, methamphetamines, opiates, cocaine, benzodiazepines, MDMA, and oxycodone collected from youth participants. Assessed at baseline and 5 months; data reported for 5-month time point
Time Frame: Baseline to 5 months
Measure: Number; unit: participants
Arm/Group | Caregiver Contingency Management + Usual Drug Court Treatment | Usual Drug Court Treatment
Number analyzed (Participants) | 18 | 13
participants | 18 | 13

2. Primary Outcome: Frequency of Substance Use and Substance-related Problems Self-reported by Youth on the Global Appraisal of Individual Needs.
Description: The GAIN Substance Frequency Scale assesses frequency of substance use over the past 90 days. Scores range from 0 (no use) to 90 (daily use). Higher scores indicate greater substance use severity.
Time Frame: Baseline, 5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregiver Contingency Management + Usual Drug Court Treatment | Usual Drug Court Treatment
Number analyzed (Participants) | 18 | 13
score on a scale
  Baseline - Days drunk or high whole day | 2.56 (6.0) | 8.03 (10.3)
  Baseline - Days of marijuana use | 4.26 (9.3) | 12.69 (13.3)
  Baseline - Days of alcohol use | 0.63 (1.63) | 2.85 (4.8)
  Month 5 - Days drunk or high whole day | 0.72 (2.4) | 4.08 (7.6)
  Month 5 - Days of marijuana use | 1.11 (3.2) | 4.54 (8.4)
  Month 5 - Days of alcohol use | 0.63 (1.8) | 1.46 (2.3)

3. Secondary Outcome: Changes From Baseline to 18 Months Post-baseline in Youth Arrests, Charges, and Convictions.
Description: Number of youth arrests, charges, and convictions measured via official arrest records.
Time Frame: Baseline to 18 months
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Changes From Baseline to 18 Months Post-baseline in Youth Delinquent Behaviors (Measured at 0, 3, 5, 6, 9, 12, and 18 Months).
Description: Frequency of delinquent behaviors self-reported by youth using the Self-Report Delinquency Scale.
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Changes From Baseline to 18 Months Post-baseline in Caregiver Reports on Youth Internalizing Symptoms and Externalizing Behaviors (Measured at 0, 1, 2, 3, 4, 5, 6, 9, 12, and 18 Months).
Description: Frequency of youth's internalizing symptoms and externalizing behaviors measured with the Child Behavior Checklist (caregiver report).
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Changes From Baseline to 18 Months Post-baseline in Youth Reports on Youth Internalizing Symptoms and Externalizing Behaviors (Measured at 0, 1, 2, 3, 4, 5, 6, 9, 12, and 18 Months).
Description: Frequency of youth's internalizing symptoms and externalizing behaviors measured with the Brief Problem Checklist (youth report).
Time Frame: Baseline to 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Changes From Baseline to Post-treatment in Caregiver Substance Use Problems.
Description: Frequency and severity of substance use problems self-reported by caregivers on the Addiction Severity Index.
Time Frame: Baseline through treatment completion, an average of 4 months
Reporting Status: Not Posted

8. Secondary Outcome: Changes From Baseline to Post-treatment in Caregiver Depressive Symptoms.
Description: Frequency and severity of depressive symptoms self-reported by caregivers on the Beck Depression Inventory.
Time Frame: Baseline through treatment completion, an average of 4 months
Reporting Status: Not Posted

9. Secondary Outcome: Changes From Baseline to Post-treatment in Therapist-Family Working Alliance (Measured at 1, 2, 3, and 4 Months, as Well as Post-treatment).
Description: Levels of alliance during treatment reported by therapists, caregivers, and youth on the Working Alliance Inventory.
Time Frame: Baseline through treatment completion, an average of 4 months
Reporting Status: Not Posted

10. Secondary Outcome: Changes From Baseline to Post-treatment in Caregiver Treatment Attendance and Activity Completion (Measured at 1, 2, 3, and 4 Months, as Well as Post-treatment).
Description: Frequency of caregiver attendance at their youth's substance use treatment sessions and completion of therapeutic activities reported by therapists on the Session Tracking Sheet.
Time Frame: Baseline through treatment completion, an average of 4 months
Reporting Status: Not Posted

11. Secondary Outcome: Changes From Baseline to the End of JDC Involvement in Caregiver Attendance at JDC Sessions.
Description: Frequency of caregiver attendance at their youth's JDC sessions reported by JDC personnel on the JDC Attendance Form.
Time Frame: Baseline through the end of JDC involvement, an average of 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Rates of Treatment Completion.
Description: Rates of youth treatment completion reported by therapists using the Treatment Termination Form.
Time Frame: Up to 4 months on average
Reporting Status: Not Posted

13. Secondary Outcome: Levels of Satisfaction With Treatment and JDC.
Description: Levels of satisfaction with substance use treatment and JDC reported by caregivers and youth on the Client Satisfaction Questionnaire.
Time Frame: Up to 4 months on average
Reporting Status: Not Posted

14. Secondary Outcome: Changes From Baseline to Post-treatment in Caregiver Perceptions of Incentive Programs.
Description: Ratings by caregivers on perceptions of incentive-based interventions as measured by the Provider Survey of Incentives.
Time Frame: Baseline through treatment completion, an average of 4 months
Reporting Status: Not Posted

15. Secondary Outcome: Changes From Baseline to 36 Months Post-baseline in Therapist and JDC Personnel Perceptions of Incentive Programs (Measured at 0, 12, 24, and 36 Months).
Description: Ratings by therapists and JDC personnel on perceptions of incentive-based interventions as measured by the Provider Survey of Incentives.
Time Frame: Baseline to 36 months
Reporting Status: Not Posted

16. Secondary Outcome: Reports at Post-treatment on Youth and Caregiver Attitudes Toward Incentive Programs.
Description: Youth and caregiver attitudes toward incentive programs as measured during qualitative interviews.
Time Frame: Up to 4 months on average
Reporting Status: Not Posted

17. Secondary Outcome: Changes From Baseline to 36 Months Post-baseline in Therapist and JDC Personnel Attitudes Toward Incentive Programs (Measured at 0, 12, 24, and 36 Months).
Description: Therapist and JDC personnel attitudes toward incentive programs as measured during qualitative interviews.
Time Frame: Baseline to 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Five months
Description: Adverse event data were collected only for adolescent participants. No adverse event data were collected for caregivers.
Groups:
- Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents): This group will receive a caregiver contingency management intervention plus the standard outpatient substance abuse treatment services provided at JDC.
  Adverse Measures are for the adolescent participants
- Usual Drug Court Treatment (Adolescents): This group will receive the standard outpatient substance abuse treatment services provided at JDC.
  Adverse Measures are for the adolescent participants
Arm/Group | Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents) | Usual Drug Court Treatment (Adolescents)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/32 | 3/21
Other Adverse Events (participants affected / at risk) | 1/32 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents) (N=32) | Usual Drug Court Treatment (Adolescents) (N=21)
Suicide attempt (Psychiatric disorders) | 3 (3) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Contingency Management + Usual Drug Court Treatment (Adolescents) (N=32) | Usual Drug Court Treatment (Adolescents) (N=21)
Emotional distress about prizes (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03051997/Prot_SAP_000.pdf